CLINICAL TRIAL: NCT00808899
Title: Neuroblastoma Protocol 2008: Therapy for Children With Advanced Stage High Risk Neuroblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Voluntarily closed and terminated by the PI due to lack of feasibility
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB2008
Record Dates: First submitted 2008-12-11; First posted 2008-12-16 (Estimated); Results first posted 2010-05-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2010-05

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — temsirolimus; Irinotecan; Cyclophosphamide; Doxorubicin; Etoposide; Cisplatin; Topotecan; Radiotherapy; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Fixed doses of IV temsirolimus concomitantly with two courses of fixed dosages of irinotecan, 2 days off, repeated daily 5 times.If initial dosages are not tolerable, subsequent patients will be given a reduced dosage of temsirolimus with irinotecan.If this dosage combination is not tolerable,irinotecan dosage will be decreased.If this dosage combination is not tolerable.Further enrollment to initial six week treatment will be terminated.Second course of irinotecan will begin on day 22, response will be determined after six weeks. Resection of primary tumor will be attempted after initial therapy.Following initial treatment children will undergo alternating courses of induction chemotherapy with cyclophosphamide,doxorubicin,etoposide,topotecan, and cisplatin.First cohort of 17 patients will receive Block 2 with temsirolimus for all three courses, weekly 2 times.If this is not tolerated subsequent patients will receive Block 2 chemotherapy with reduced dosages of temsirolimus.
  Interventions: Drug: Temsirolimus; Drug: Irinotecan; Procedure: Surgical Resection of Primary Tumor; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Cisplatin; Drug: Topotecan; Procedure: PBSC; Radiation: Radiation Therapy; Drug: 13-cis-retinoic acid

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus
Drug: Irinotecan — Irinotecan
Procedure: Surgical Resection of Primary Tumor — Surgical Resection of Primary Tumor
Drug: Cyclophosphamide — Cyclophosphamide
Drug: Doxorubicin — Doxorubicin
Drug: Etoposide — Etoposide
Drug: Cisplatin — Cisplatin
Drug: Topotecan — Topotecan
Procedure: PBSC — Peripheral Blood Stem Cell Harvest
Radiation: Radiation Therapy — Radiation Therapy
Drug: 13-cis-retinoic acid — 13-cis-retinoic acid

SUMMARY:
A Phase II study of temsirolimus in combination with standard chemotherapy (irinotecan; cyclophosphamide, doxorubicin and etoposide (CAE); cisplatin and etoposide (HiPE) and topotecan (TPT) followed by and additional six courses of induction chemotherapy and then intensification with autologous hematopoietic stem cell transplantation. The first five courses of induction chemotherapy will also evaluate the feasibility of combining weekly temsirolimus with these standard chemotherapy combinations. This will be followed by 16 months of oral maintenance therapy with eight months of 13-cis-retinoic acid and then eight months of oral topotecan.

DETAILED DESCRIPTION:
All children will receive fixed doses of intravenous temsirolimus (50 mg/m2 weekly 6 times ) concomitantly with two courses of fixed dosages of irinotecan (20 mg/m2 intravenously daily 5 times ,2 days off, repeated daily 5 times .If these initial dosages are not tolerable then subsequent patients will be given a reduced dosage of temsirolimus (25 mg/m2 weekly 6 times) with 20 mg/m2 of irinotecan.If this dosage combination is not tolerable, the irinotecan dosage will be decreased to 15 mg/m2 .If this dosage combination is not tolerable then further enrollment to the initial six week treatment will be terminated.The second course of irinotecan will begin on day 22 and response will be determined after six weeks (two courses). Resection of primary tumor will be attempted after this initial therapy, whenever possible.

Following initial treatment children will undergo alternating courses of induction chemotherapy with cyclophosphamide, doxorubicin, etoposide, topotecan, and cisplatin (Block 2). The first cohort of 17 patients will receive Block 2 with temsirolimus (50mg/m2) for all three courses, weekly 2 times. If this is not tolerated subsequent patients will receive Block 2 chemotherapy with reduced dosages of temsirolimus (25mg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Patients <18 years old with newly diagnosed, advanced stage, high-risk neuroblastoma defined as one of the following:

  * Children < 1 yo with International Neuroblastoma Staging System (INSS) stage 2a, 2b, 3, 4 or 4S disease and MYCN amplification (>10 copies, or greater than four-fold increase in MYCN signal as compared to reference signal)
  * INSS 2a or 2b disease and MYCN amplification, regardless of age or additional biologic features
  * INSS stage 3 and:

    1. MYCN amplification (>10 copies, or greater than four-fold increase in MYCN signal as compared to reference signal, regardless of age or additional biologic features
    2. Age > 18 mo (> 547 days) with unfavorable pathology, regardless of MYCN status
  * INSS stage 4 and:

    1. MYCN amplification, regardless of age or additional biologic features
    2. Age > 18 months (> 547 days) regardless of biologic features
    3. Age 12 - 18 months (365 - 547 days) with any of the following three unfavorable biologic features (MYCN amplification, unfavorable pathology and/or DNA index =1) or any biologic feature that is indeterminant/unknown
  * Children less than or equal to 365 days initially diagnosed with: INSS stage 1, 2, 4S who progressed to a stage 4 without interval chemotherapy.
* Histologic proof of neuroblastoma or positive bone marrow for tumor cells with increased urine catecholamines.
* Adequate renal and hepatic function (serum creatinine <3 x upper limit of normal for age, (AST) aspartate aminotransferase < 3 x upper limit of normal).
* No prior therapy, unless an emergency situation requires local tumor treatment (discuss with PI)
* Written, informed consent according to institutional guidelines

Exclusion Criteria:

* Any evidence, as judged by the investigator, of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* Pregnant or breast feeding (women of child-bearing potential).
* Children with INSS 4 disease, age <12 months with all 3 favorable biologic features (non-amplified MYCN, favorable pathology and DNA index >1).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Furman, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four patients were recruited from December, 2008 through April, 2009. The study was suspended July, 2009 because of the publication of a new standard of care in treatment for patients with high-risk neuroblastoma.
Groups:
- Temsirolimus With Irinotecan: Participants enrolled in the Temsiolimus and Irinotecan group were high-risk neuroblastoma patients.
Period: Overall Study
Arm/Group | Temsirolimus With Irinotecan
Started | 4
Completed | 0
Not Completed | 4
Not completed — Death | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Temsirolimus With Irinotecan
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.5 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Plus Partial Response
Description: The objective was to measure the efficacy and feasability of Temsirolimus and Irinotecan as measured by the objective response rate and toxicity rate.
Time Frame: 10 years
Population: The population consisted of patients eligible for enrollment onto the NB2008 protocol.
Arm/Group | Temsirolimus With Irinotecan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Temsirolimus With Irinotecan
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus With Irinotecan (N=4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory, Lung (Pulmonary Hemorrhage) (Blood and lymphatic system disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus With Irinotecan (N=4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (2)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (4)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 4 (16)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (2)
Hemoglobin (Blood and lymphatic system disorders) | 4 (25)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 3 (7)
Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related, Wound (Infections and infestations) | 1 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (25)
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (25)
Pain, Abdomen NOS, Bone, Extremity, Limb, Oral Cavity (General disorders) | 4 (5)
Phosphate, serum-low (hypophosphatemia) (General disorders) | 4 (11)
Platelets (Blood and lymphatic system disorders) | 4 (22)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (10)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (3)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
NB2008 was closed because of the publication of a new standard of care for treating high-risk neuroblastoma.At the time of closure, NB2008 had enrolled only 4 patients, which was an insufficient number of patients to answer the primary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes